CLINICAL TRIAL: NCT04380480
Title: A Prospective, Phase II Study of Percutaneous Endoscopic Gastrostomy Before Definitive Concurrent Chemoradiation Therapy in Patients With Esophageal Squamous Cell Carcinoma
Brief Title: Percutaneous Endoscopic Gastrostomy Before Definitive Concurrent Chemoradiation Therapy for Esophageal Squamous Cell Carcinoma
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Sun Yat-sen University (Other)
Responsible Party: Principal Investigator, Hui Liu, Professor, Sun Yat-sen University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: GASTO-1059
Record Dates: First submitted 2020-03-21; First posted 2020-05-08 (Actual); Last update posted 2023-01-11 (Actual); Status verified 2023-01

CONDITIONS: Esophageal Squamous Cell Carcinoma
Keywords: esophageal squamous cell carcinoma; percutaneous endoscopic gastrostomy; concurrent chemoradiotherapy; enteral nutrition support
MeSH Terms: conditions — Esophageal Squamous Cell Carcinoma

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Experiment (Experimental): One or two weeks before CCRT, all patients will undergo a percutaneous endoscopic gastrostomy (PEG) to be administered enteral nutrition support(30-35 kcal/kg of energy, 1.2-1.5g/kg of protein and electrolyte supplementation each day). Nutritional supplements will be administered till 1 month after CCRT.
  All patients will receive definitive radiotherapy combined with three cycles of S-1 (40mg/2, BID, po) on D1-14, D22-35, D43-56.
  Interventions: Combination Product: Concurrent chemoradiotherapy combined with enteral feeding by percutaneous endoscopic gastrostomy

INTERVENTIONS:
Combination Product: Concurrent chemoradiotherapy combined with enteral feeding by percutaneous endoscopic gastrostomy — One or two weeks before CCRT, all patients will undergo a percutaneous endoscopic gastrostomy (PEG) to be administered enteral nutrition support(30-35 kcal/kg of energy, 1.2-1.5g/kg of protein and electrolyte supplementation each day). Nutritional supplements will be administered till 1 month after CCRT.
  All patients will receive definitive radiotherapy combined with three cycles of S-1 (40mg/2, BID, po) on D1-14, D22-35, D43-56.

SUMMARY:
This Phase II randomized study is to determine the efficacy of percutaneous endoscopic gastrostomy before definitive concurrent chemoradiotherapy (CCRT) in Patients with Esophageal Squamous Cell Carcinoma(ESCC) by assessing their weight, nutritional status, performance status and treatment response.

DETAILED DESCRIPTION:
This Phase II randomized study is to determine the efficacy of percutaneous endoscopic gastrostomy before definitive concurrent chemoradiotherapy (CCRT) in Patients with Esophageal Squamous Cell Carcinoma(ESCC) by assessing their weight, nutritional status, performance status and treatment response.

All patients will receive definitive radiotherapy combined with three cycles of S-1 (40mg/2, BID, po) on D1-14, D22-35, D43-56. The primary endpoint is percentage of recent weight loss at the end of CCRT. The secondary endpoints are nutrition status, objective response rate, overall survival, toxicity and intestinal flora changes in blood, urine and stool specimens.

ELIGIBILITY:
Inclusion Criteria:

* Histologically confirmed esophageal squamous cell carcinoma
* Patients have measurable or evaluable lesions based on the Response Evaluation Criteria in Solid Tumors (RECIST) criteria.
* Eastern Cooperative Oncology Group (ECOG) performance status 0-1.
* Estimated life expectancy of at least 6 months
* No contraindications for chemotherapy or radiotherapy
* Patients and their family signed the informed consents

Exclusion Criteria:

* Severe gastrointestinal impairment or enteral nutrition intolerance
* Severe vomiting, gastrointestinal bleeding or intestinal obstruction
* Severe malnutrition
* Patients with contraindications for percutaneous endoscopic gastrostomy, including uncorrected coagulopathy or thrombocytopenia, varices caused by portal hypertension, or other gastric diseases
* Not suitable for this study judged by researchers

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 63 (Actual)
Dates: Start 2020-02-01 (Actual); Primary Completion 2022-03-15 (Actual); Study Completion 2022-03-15 (Actual)

PRIMARY OUTCOMES:
Percentage of Recent Weight Loss | From baseline until the end of concurrent chemoradiotherapy, an average of 8 weeks

SECONDARY OUTCOMES:
Change in nutrition status assessed by blood test | 1 year
  Change in nutrition status will be assessed by hemoglobin, serum albumin, pre-albumin test. The patient-generated subjective global assessment will also be used to measure patients' nutrition status
Quality of life measured by WHO Quality of Life-100 questionnaire | 1 year
Rate of grade 3-4 radiation esophagitis | 1 year
Rate of grade 3-4 radiation pneumonitis， | 1 year
Rate of grade 3-4 bone marrow suppression | 1 year
Objective response rate | 2 months
Overall survival | 3 years
Changes of participants' intestinal flora assessed by blood, urine and stool test | 1 year

CONTACTS AND LOCATIONS:
Overall Officials: Hui Liu, Ph.D, Principal Investigator — Sun Yat-sen University
Locations (1):
- Hui Liu, Guangzhou, Guangdong, China

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Torre LA, Bray F, Siegel RL, Ferlay J, Lortet-Tieulent J, Jemal A. Global cancer statistics, 2012. CA Cancer J Clin. 2015 Mar;65(2):87-108. doi: 10.3322/caac.21262. Epub 2015 Feb 4. PMID 25651787
- [Background] Cooper JS, Guo MD, Herskovic A, Macdonald JS, Martenson JA Jr, Al-Sarraf M, Byhardt R, Russell AH, Beitler JJ, Spencer S, Asbell SO, Graham MV, Leichman LL. Chemoradiotherapy of locally advanced esophageal cancer: long-term follow-up of a prospective randomized trial (RTOG 85-01). Radiation Therapy Oncology Group. JAMA. 1999 May 5;281(17):1623-7. doi: 10.1001/jama.281.17.1623. PMID 10235156
- [Background] Bozzetti F, Mariani L, Lo Vullo S; SCRINIO Working Group; Amerio ML, Biffi R, Caccialanza G, Capuano G, Correja I, Cozzaglio L, Di Leo A, Di Cosmo L, Finocchiaro C, Gavazzi C, Giannoni A, Magnanini P, Mantovani G, Pellegrini M, Rovera L, Sandri G, Tinivella M, Vigevani E. The nutritional risk in oncology: a study of 1,453 cancer outpatients. Support Care Cancer. 2012 Aug;20(8):1919-28. doi: 10.1007/s00520-012-1387-x. Erratum In: Support Care Cancer. 2012 Aug;20(8):1929. Capuano, Giovanni [corrected to Capuano, Giorgio]. PMID 22314972
- [Background] Clavier JB, Antoni D, Atlani D, Ben Abdelghani M, Schumacher C, Dufour P, Kurtz JE, Noel G. Baseline nutritional status is prognostic factor after definitive radiochemotherapy for esophageal cancer. Dis Esophagus. 2014 Aug;27(6):560-7. doi: 10.1111/j.1442-2050.2012.01441.x. Epub 2012 Oct 26. PMID 23106980
- [Background] Ma L, Luo GY, Ren YF, Qiu B, Yang H, Xie CX, Liu SR, Liu SL, Chen ZL, Li Q, Fu JH, Liu MZ, Hu YH, Ye WF, Liu H. Concurrent chemoradiotherapy combined with enteral nutrition support: a radical treatment strategy for esophageal squamous cell carcinoma patients with malignant fistulae. Chin J Cancer. 2017 Jan 11;36(1):8. doi: 10.1186/s40880-016-0171-6. PMID 28077159
- [Background] Birnstein E, Schattner M. Nutritional Support in Esophagogastric Cancers. Surg Oncol Clin N Am. 2017 Apr;26(2):325-333. doi: 10.1016/j.soc.2016.10.003. Epub 2017 Feb 9. PMID 28279472
- [Background] Yu FJ, Shih HY, Wu CY, Chuang YS, Lee JY, Li HP, Fang PT, Tsai DL, Chou SH, Wu IC. Enteral nutrition and quality of life in patients undergoing chemoradiotherapy for esophageal carcinoma: a comparison of nasogastric tube, esophageal stent, and ostomy tube feeding. Gastrointest Endosc. 2018 Jul;88(1):21-31.e4. doi: 10.1016/j.gie.2017.11.030. Epub 2017 Dec 7. PMID 29225081
- [Background] Lin CH, Liu NJ, Lee CS, Tang JH, Wei KL, Yang C, Sung KF, Cheng CL, Chiu CT, Chen PC. Nasogastric feeding tube placement in patients with esophageal cancer: application of ultrathin transnasal endoscopy. Gastrointest Endosc. 2006 Jul;64(1):104-7. doi: 10.1016/j.gie.2005.12.036. PMID 16813813
- [Background] Margolis M, Alexander P, Trachiotis GD, Gharagozloo F, Lipman T. Percutaneous endoscopic gastrostomy before multimodality therapy in patients with esophageal cancer. Ann Thorac Surg. 2003 Nov;76(5):1694-7; discussion 1697-8. doi: 10.1016/s0003-4975(02)04890-7. PMID 14602314
- [Background] Sofue K, Takeuchi Y, Tsurusaki M, Shibamoto K, Sakamoto N, Kitajima K, Sone M, Sugimura K, Arai Y. Value of Percutaneous Radiologic Gastrostomy for Patients with Advanced Esophageal Cancer. Ann Surg Oncol. 2016 Oct;23(11):3623-3631. doi: 10.1245/s10434-016-5276-2. Epub 2016 May 17. PMID 27188297